CLINICAL TRIAL: NCT05270486
Title: Safety and Efficacy of Electromagnetic Navigation System Assisted Percutaneous Endoscopic Lumbar Decompression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Remacle Thibault, Principal Investigator, MD, PhD, Neurosurgeon, Centre Hospitalier Régional de la Citadelle
Other Study IDs: EM Assisted TELD
Record Dates: First submitted 2022-01-29; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Cervical Foraminal Stenosis; Cervical Disc Herniation
Keywords: electromagnetic navigation; herniated disc; transforaminal endoscopic lumbar discectomy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group A: group A undergoing TELD (transforaminal endoscopic lumbar discectomy) with electromagnetic navigation system
  Interventions: Procedure: Electromagnetic navigation system
- Group B: group B undergoing TELD with X-ray fluoroscopy (gold standard)

INTERVENTIONS:
Procedure: Electromagnetic navigation system — The aim of this study is to assess the safety and efficacy of TELD assisted by electromagnetic navigation for treating lumbar disc herniation (LDH).
  Groups: Group A

SUMMARY:
There is a shallow learning curve with TELD (transforaminal endoscopic lumbar discectomy). The aim of this study is to assess the safety and efficacy of TELD assisted by electromagnetic navigation for treating lumbar disc herniation (LDH).

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 and ≤80 years;
2. typical clinical symptoms and consistent imaging evidence of mono-radiculopathy LDH; or single level LSS combined with disc herniation
3. recalcitrant pain despite proper conservative therapy (including analgesics, NSAIDs, corticoids infusion under CT guidance and physical therapy) for at least 3 months before surgery and/or neurological deficit in the territory of the irritated nerve root
4. VAS pain ≥ 6/10
5. Absence of significant instability;

Exclusion Criteria:

1. serious underlying disease or mental illnesses
2. severe central stenosis, cauda equina syndrome, spinal instability, active infection, and serious calcified fragments
3. previous lumbar treatment with spinal surgery, ozone intervention, or radiofrequency ablation
4. unwilling or unable to participate in treatment and complete follow-up
5. Multi-level disc pathology
6. MRC paresis <4/5
7. Pregnancy
8. participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 consecutive patients, group A undergoing TELD with electromagnetic navigation system vs. group B undergoing TELD with X-ray fluoroscopy (gold standard). Parameters: gender, age, body mass index, neurological examination, comorbidities (diabetes, AHT, depression, smoking, work status, other joint problems), recurrence of disc herniation, follow-up time, pain evaluation on the day before surgery (numerical rating scale), herniation level, type of herniation (disc protrusion, disc prolapsed, disc extrusion or sequestered disc), duration of preoperative back pain/leg pain, use of analgesics (type and duration), preoperative Roland-Morris disability questionnaire, preoperative Oswestry Disability Index.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | Preoperatively. 6 weeks, 3 months, 6 months and 12 months post-operatively
  0% to 20%: minimal disability: The patient can cope with most living activities. Usually no treatment is indicated apart from advice on lifting sitting and exercise. 21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means. 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation. 61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required. 81%-100%: These patients are either bed-bound or exaggerating their symptoms.
Change in Roland Morris Disability Questionnaire (RMDQ) | Preoperatively. 6 weeks, 3 months, 6 months and 12 months post-operatively
  This is a 24 item questionnaire. The patient is asked to tick a statement when it applies to him that specific day, this makes it possible to follow changes in time. The end score is the sum of the ticked boxes. The score ranges from 0 (no disability) to 24 (max. disability)

SECONDARY OUTCOMES:
Back Pain Numerical Rating Score (BPNRS) | Preoperatively. 6 weeks, 3 months, 6 months and 12 months post-operatively
  Patient is asked to rate his pain between 11 points (0-11; 0=no pain and 10=worst pain imaginable)
Leg Pain Numerical Rating Score (LPNRS) | Preoperatively. 6 weeks, 3 months, 6 months and 12 months post-operatively
  Patient is asked to rate his pain between 11 points (0-11; 0=no pain and 10=worst pain imaginable)
Modified MacNab Criteria | Preoperatively. 6 weeks, 3 months, 6 months and 12 months post-operatively
  Patient is asked about his well being and has to choose between:
  Excellent: No pain, No restriction of mobility, Return to normal work and level of activity Good: Occasional nonradicular pain, Relief of presenting symptoms, Able to return to modified work Fair: Some improved functional capacity, Still handicapped and/or unemployed Poor: Continued objective symptoms of root involvement, Additional operative intervention needed at index level irrespective of length of postoperative follow-up

IPD SHARING:
Plan to Share IPD: Undecided